CLINICAL TRIAL: NCT05356988
Title: Health and Energy Through Active Living Every Day After Cancer Intervention for Cancer Survivors
Acronym: HEALED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CPS3HEALED
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Cognitive Decline; Fatigue; Sleep; Anxiety; Depression
Keywords: cancer; physical activity; sedentary behavior
MeSH Terms: conditions — Cognitive Dysfunction; Fatigue; Anxiety Disorders; Depression; Neoplasms; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The intervention group will have access for one year to a website to help increase aerobic and strength training activities. The control group will have access for one year to a website to help improve balance and flexibility. At the end of the one-year study, each group will get access to the opposite website.
Masking Description: Investigator will not be involved in randomization, but given the obvious differences in treatment vs. control, participants, investigator, and assessors will be aware of assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Group (Experimental): Physical activity (PA) group participants will receive behavioral nudge e-mails with links to a web-based platform which will provide: physical activity information, at-home exercise demonstrations/videos for survivors of all fitness levels, articles, blog posts, physical activity/sitting recommendations, a space for goal setting, a platform for physical activity tracking, a discussion board, automatic syncing of their Fitbit to the leaderboard, etc.
  Interventions: Behavioral: Physical activity experiment
- Balance and Flexibility Group (Active Comparator): The static Balance and Flexibility (BF) website will include infographics, videos, and articles for participants to view at their leisure. They will receive access to the HEALED website at the end of the 12-month intervention period.
  Interventions: Behavioral: Balance and flexibility control

INTERVENTIONS:
Behavioral: Physical activity experiment — The Physical Activity (PA) group will have access for one year to the PA website to help increase aerobic and strength training activities.
  Arms: Physical Activity Group
Behavioral: Balance and flexibility control — The static Balance and Flexibility (BF) website will include infographics, videos, and articles for participants to view at their leisure around stretching and balance exercises.
  Arms: Balance and Flexibility Group

SUMMARY:
The purpose of the Health and Energy through Active Living Every Day (HEALED) intervention, is to examine the effect of a web-based intervention on changes in device-measured physical activity (light and moderate-to-vigorous intensity aerobic) and sedentary behavior. The purpose of this study is intended for survivors of a cancer with a 5-year survival (at Stage I, II, and III) of at least 45% that has a strong level of evidence for association with physical inactivity according to the 2018 PA Guidelines Advisory Committee Report (breast, colon, endometrium, kidney, bladder, multiple myeloma). In line with social cognitive theory behavior change techniques, participants will be provided information and skills necessary to be more physically active and less sedentary after a cancer diagnosis. New materials will be disseminated biweekly through a website open only to participants, and include at-home exercise demonstration videos, research news, discussion boards, success stories, infographics for exercise recommendations, etc.

DETAILED DESCRIPTION:
By 2026, there will be approximately 20.3 million cancer survivors in the U.S., and this population is expected to grow with improved cancer survival rates. Cancer survivors experience a myriad of side effects following treatment, including fatigue, decreased muscle mass, balance issues, decreased cognitive function, and an increased risk of comorbidities. Observational studies and randomized controlled trials suggest that physical activity (PA) is a safe and effective non-pharmacologic option for improving some of these side effects. Despite the evidence, it is estimated that at least 75% of cancer survivors do not meet PA guidelines. Interventions tailored for survivors may increase PA, but there are gaps in the literature regarding the most effective methods. Further, there are several cancers associated with physical inactivity, but most PA interventions focus on breast cancer. Additionally, many existing interventions require in-person meetings, are very resource-intensive, and may not be sustainable. Most physical activity interventions focus on the promotion of moderate-vigorous PA, ignoring the importance of decreased sedentary time and increased light PA. Accordingly, it is imperative to create more sustainable, broad-reaching PA and sedentary behavior interventions that are intended for survivors of various physical inactivity-associated cancers. The proposed one-year study will be a two-arm, randomized control intervention embedded within the Cancer Prevention Study-3 (CPS-3), a prospective cohort study of cancer incidence and mortality initiated by the American Cancer Society. The proposed Health and Energy through Active Living Every Day (HEALED) intervention is intended for survivors of a cancer with an expected 5-year survival (at Stage I, II or III) of at least 45% that has a strong level of evidence for association with physical inactivity according to the 2018 PA Guidelines Advisory Committee Report (breast, colon, endometrium, kidney, multiple myeloma, and bladder). In line with social cognitive theory behavior change techniques, participants will be provided information and skills necessary to be more physically active and less sedentary after a cancer diagnosis. Materials and tools will be updated monthly through a secure website open only to participants, and include: at-home exercise demonstration videos, steps leaderboards, goal setting tools, Fitbit self-monitoring and syncing capabilities, discussion boards, success stories, infographics for exercise recommendations, etc. This intervention will add to the very minimal evidence base for PA interventions for diverse cancer survivors in a sustainable, broad-reaching manner. Further, the data resulting from this study will provide insight towards promotion of the "time-use" approach, which focuses on all of the movement behaviors (including sedentary time, light intensity physical activity, and moderate-to-vigorous physical activity), which has not yet been used in interventions for survivors.

ELIGIBILITY:
Inclusion Criteria:

* Are a survivor of Stage I - III breast, colon, endometrium, kidney, or bladder cancer, or of multiple myeloma (verified through medical record abstraction/tumor tissue or state registry, to which participants have already consented)
* Are a part of the CPS-3 Portal (this also implies that an email address is on file and an English survey response)
* Must have a physical, continental US street address where they can receive shipments for 12 months.
* Have access to a working smartphone or tablet
* Are not currently pregnant
* Exercise less 300 minutes per week
* Did not register for HEALED Study pilot (n = 99; conducted in 2019, published in 2021; Appendix 11, AM12_IRB00059007 approved in February 2019)
* Are able to walk assisted

Exclusion Criteria:

* A doctor has recommended that they avoid moderate or vigorous exercise, or limit walking
* Have received any of the following treatments for their cancer diagnosis in the last 6 months: Surgery to remove the cancer, chemotherapy, radiation therapy, or immunotherapy.
* Have major planned surgery in the next 12 months

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Sedentary time | 12 months
  Device-measured sedentary time with research-grade accelerometer
Physical activity | 12 months
  Device-measured light, moderate, vigorous intensity physical activity with research-grade accelerometer and Fitbit.

SECONDARY OUTCOMES:
PROMIS Sleep Disturbance | 12 months
  5-item questionnaire measuring self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep problems during waking hours within the past seven days.
CPS-3 Fatigue Questions | 12 months
  A 5-item Likert scale measuring fatigue, lack of energy and general tiredness within the past month.
PROMIS Global Mental and Physical Health | 12 months
  Instrument consists of ten global health items that represent five core PROMIS domains (physical function, pain, fatigue, emotional distress, social health). Four items are used to assess global physical health. Four items are used to assess global mental health, all of which are administered using five-category response scales. Higher scores indicate better mental/physical health.
Emotional Distress-Anxiety | 12 months
  A PROMIS assessment of 8-items on the pure domain of anxiety in individuals age 18 and older. High scores indicate higher anxiety symptom severity.
Emotional Distress-Depression | 12 months
  A PROMIS assessment of 7-items on the pure domain of depression in individuals age 18 and older. High scores indicate higher depression symptom severity.
PROMIS Cognitive Function | 12 months
  This item bank assesses patient-perceived cognitive deficits. Facets include mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in cognitive functions. Higher scores indicate higher cognitive funciton.
30 second sit-stand test | 12 months
  Video-administered, self-reported sit-stand test (validity study: https://pubmed.ncbi.nlm.nih.gov/34797895/)

CONTACTS AND LOCATIONS:
Locations (1):
- American Cancer Society (virtual recruitment and study), Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rees-Punia E, Leach CR, Westmaas JL, Dempsey LF, Roberts AM, Nocera JR, Patel AV. Pilot Randomized Controlled Trial of Feasibility, Acceptability, and Preliminary Efficacy of a Web-Based Physical Activity and Sedentary Time Intervention for Survivors of Physical Inactivity-Related Cancers. Int J Behav Med. 2022 Apr;29(2):220-229. doi: 10.1007/s12529-021-09999-5. Epub 2021 May 6. PMID 33954891
- [Derived] Rees-Punia E, Masters M, Whalen S, Hartman SJ, Sullivan K, Westmaas JL, Teras LR, Patel AV. Digital intervention for increasing physical activity and reducing sedentary behaviour in cancer survivors: a trial within the Cancer Prevention Study-3 cohort. Br J Sports Med. 2025 Jul 31;59(16):1143-1150. doi: 10.1136/bjsports-2024-109332. PMID 40461052

DOCUMENTS (1):
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT05356988/ICF_000.pdf